CLINICAL TRIAL: NCT02823795
Title: The Supporting Patient Activation in Transition to Home (sPATH) Intervention - a Study Protocol of Randomized Controlled Trial
Brief Title: The Supporting Patient Activation in Transition to Home Intervention
Acronym: [sPATH]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Vårdalstiftelsen (Unknown); Forte (Industry)
Responsible Party: Principal Investigator, Mirjam Ekstedt, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C751231003; Dnr 2014-0026 (Other Grant/Funding Number: Vårdalsstiftelsen); Dnr 2014-4948 (Other Grant/Funding Number: Forte)
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Medication Adherence; Self-care; Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Patient participation; Empowerment; Medication management; Symptom management; Self determination theory; Motivational Interviewing
MeSH Terms: conditions — Medication Adherence; Heart Failure; Pulmonary Disease, Chronic Obstructive; Patient Participation; Empowerment | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sPATH (Experimental): Motivational Interviewing in five sessions post hospital discharge
  Interventions: Behavioral: Motivational Interviewing
- Control (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Motivational Interviewing — Patients will get motivational interviewing sessions by a patient activation coach (medical social workers and/or nurses trained in motivational interviewing and in the intervention) in five post hospital discharge sessions (whereof one face-to-face, four by phone) aiming to increase patient motivation to become active in self-management (medication management, care plan/follow-up, symptoms/signs of worsening condition, contacts with health care provider).
  Arms: sPATH

SUMMARY:
This study evaluates if motivational interviewing sessions aiming to motivate recently discharged patients with either chronic obstructive pulmonary disease or congestive heart failure to be active in post-discharge self-management can reduce re-hospitalization rates.

DETAILED DESCRIPTION:
Included patients transition to home will be bridged through a telephone-call from a patient activation coach two days post-discharge. The patients will thereafter get motivational interviewing sessions by the same patient activation coach with the the goal that the patients are motivated to the knowledge, skills and confidence needed to manage the four main activity areas: 1) medication management; 2) adhere to care plan/ follow-up visits according to the discharge plan; 3) recognize indications (symptoms/signs) that the condition is worsening and how to respond; and 4) contact and manage relations/encounters with health care providers. Patients in control group will receive standard care, i.e. discharge and follow-up as in normal procedures. The investigators will use a randomization in permuted blocks of 10 intervention patients and 10 control patients included. To test the hypothesis that the re-hospitalizations rate is 15 % lower in the intervention group compared to the control group 242 patients (121 per group) are needed for power of 80% with the level of significance set to 5 % using two-sided chi-square.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with chronic obstructive pulmonary disease or congestive heart failure admitted at a short-term medical ward and who are living in their private home.

Exclusion Criteria:

* Diagnoses of dementia or cognitive impairment, and need of interpreter to participate in conversations.

The exclusion criteria are related to the patients' possibilities to participate in the motivational interviewing sessions by phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Re-hospitalization | 90 days
  Registry data from the Swedish Register for Health Care Encounters

SECONDARY OUTCOMES:
Healthcare usage | 30, 90 and 180 days
  Registry data from the Swedish Register for Health Care Encounters: re-hospitalization at 30 and 180 days. Emergency room and primary care visits at 30, 90 and 180 days
Medication adherence | 30, 90 and 180 days
  Patient reported data using the Morisky Medication Adherence Scale, 8 items, and registry data using medicine data from the Swedish Prescribed Drug Registry
Patient activation | 30, 90 and 180 days
  Patient reported data using the Patient Activation Measure, 13 item
Health related quality of life | 30, 90 and 180 days
  Patient reported data using the EQ-5D-5L
Basic Psychological Needs | 30, 90 and 180 days
  Patient reported data using the the Basic Psychological Need Satisfaction & Frustration Scale, 18 items
Depression | 30, 90 and 180 days
  Patient reported data using PHQ-9 (Patient Health Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Ekstedt, Professor, Principal Investigator — LIME, Karolinska Institutet
Locations (2):
- Sweden (2):
  - Akutkliniken, Karolinska University Hospital, Huddinge
  - Karolinska Universitetssjukhuset, Lung- Allergikliniken, Huddinge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaltenbrunner M, Flink M, Brandberg C, Hellstrom A, Ekstedt M. Motivational interviewing for reducing rehospitalisation and improving patient activation among patients with heart failure or chronic obstructive pulmonary disease: a randomised controlled trial. BMJ Open. 2025 Apr 14;15(4):e081931. doi: 10.1136/bmjopen-2023-081931. PMID 40228854
- [Derived] Adelsjo I, Lehnbom EC, Hellstrom A, Nilsson L, Flink M, Ekstedt M. The impact of discharge letter content on unplanned hospital readmissions within 30 and 90 days in older adults with chronic illness - a mixed methods study. BMC Geriatr. 2024 Jul 10;24(1):591. doi: 10.1186/s12877-024-05172-1. PMID 38987669
- [Derived] Brandberg C, Ekstedt M, Flink M. Self-management challenges following hospital discharge for patients with multimorbidity: a longitudinal qualitative study of a motivational interviewing intervention. BMJ Open. 2021 Jul 30;11(7):e046896. doi: 10.1136/bmjopen-2020-046896. PMID 34330857
- [Derived] Flink M, Brandberg C, Ekstedt M. Why patients decline participation in an intervention to reduce re-hospitalization through patient activation: whom are we missing? Trials. 2019 Jan 25;20(1):82. doi: 10.1186/s13063-019-3187-9. PMID 30683140
- [Derived] Flink M, Lindblad M, Frykholm O, Kneck A, Nilsen P, Arestedt K, Ekstedt M. The Supporting Patient Activation in Transition to Home (sPATH) intervention: a study protocol of a randomised controlled trial using motivational interviewing to decrease re-hospitalisation for patients with COPD or heart failure. BMJ Open. 2017 Jul 10;7(7):e014178. doi: 10.1136/bmjopen-2016-014178. PMID 28698319